CLINICAL TRIAL: NCT03845387
Title: A Phase II Clinical Study of KDT-3594 in Patients With Early Parkinson's Disease.
Brief Title: A Clinical Study of KDT-3594 in Patients With Early Parkinson's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KDT1201
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KDT-3594 (Experimental)
  Interventions: Drug: KDT-3594
- Pramipexole (Other): Reference drug
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: KDT-3594 — oral administration, dose titration
  Arms: KDT-3594
Drug: Pramipexole — ER formulation, oral administration, dose titration
  Arms: Pramipexole

SUMMARY:
Objective of this study is to investigate the efficacy, safety and pharmacokinetics of KDT-3594 in patients with early Parkinson's disease without a concomitant medication of L-dopa.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients
* Patients who are diagnosed with Parkinson's disease according to UK Parkinson's Disease society brain bank clinical diagnostic criteria
* Patients with Parkinson's disease in Stages 1 to 3 on the Modified Hoehn and Yahr Scale

Exclusion Criteria:

* Patients who are suspected any parkinsonism except for idiopathic Parkinson's disease
* Patients who underwent neurosurgical treatment (stereotaxic destruction, deep brain stimulation etc.) for PD, or patients for whom surgical treatment is scheduled during the study
* Patients with a complication of obvious dementia, or patients with Mini-Mental State Examination (MMSE) score < 24 points

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score | 12 weeks
  Change from baseline (Week 0) in MDS-UPDRS total score

SECONDARY OUTCOMES:
Change in Parkinson's Disease Questionnaire-39 (PDQ-39) score | 12 weeks
  Change from baseline (Week 0) in PDQ-39 summary index score
Change in Parkinson's Disease Sleep Scale-2 (PDSS-2) score | 12 weeks
  Change from baseline (Week 0) in PDSS-2 total score

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Koshihara, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan